CLINICAL TRIAL: NCT05584293
Title: DIABASE; Diabetes Mellitus Registry in Second Care
Acronym: DIABASE
Status: Recruiting | Type: Observational
Sponsor: Ziekenhuisgroep Twente (Other)
Collaborators: University of Twente (Other)
Responsible Party: Sponsor
Other Study IDs: ZGT20-40; W20.197 (Other: Medical Research Ethics Committees United)
Record Dates: First submitted 2022-10-13; First posted 2022-10-18 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to examine real world data from medical devices and clinical outcome from diabetes mellitus patients to gain the necessary insights to be able to improve individual patient care by building a registry.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 or type 2 diabetes
* Patients aged 18 years or older
* Patients visiting the outpatient clinic internal medicine in the ZGT Hospital
* Written informed consent

Exclusion Criteria:

* Severe general diseases or mental disorders making the participation in the study impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients with type 1 or type 2 diabetes mellitus.
  Patients are recruited at the outpatient clinic of internal medicine, diabetes clinic.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-09-11 (Actual); Primary Completion 2050-12-31 (Estimated); Study Completion 2060-12-31 (Estimated)

PRIMARY OUTCOMES:
Real world data from medical devices and clinical outcome in a registry | 0-30 years
  Examine real world data from medical devices and clinical outcome in a registry to gain the necessary insights to be able to improve individual patient care

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuisgroep Twente, Almelo, Overijssel, Netherlands

REFERENCES:
- [Derived] Urgert T, Kappert KDR, Veldhuis A, Geerdink J, van Beijnum BJF, Laverman GD. DIABASE: an automatically filled single-centre registry of diabetes mellitus in the Netherlands, combining clinical data with real-world longitudinal wearable device data-a study protocol. BMJ Open. 2025 Oct 13;15(10):e096888. doi: 10.1136/bmjopen-2024-096888. PMID 41083304
- [Derived] den Braber N, Braem CIR, Vollenbroek-Hutten MMR, Hermens HJ, Urgert T, Yavuz US, Veltink PH, Laverman GD. Consequences of Data Loss on Clinical Decision-Making in Continuous Glucose Monitoring: Retrospective Cohort Study. Interact J Med Res. 2024 Jul 31;13:e50849. doi: 10.2196/50849. PMID 39083801